CLINICAL TRIAL: NCT04856527
Title: The Motor Control Consequences of Excessive Physical Therapist Support in Individuals With Stroke
Brief Title: Motor Control Physical Therapist Support Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: TriHealth Inc. (Other)
Responsible Party: Principal Investigator, Sarah Schwab, Principal Investigator, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2020-1072
Record Dates: First submitted 2021-04-14; First posted 2021-04-23 (Actual); Results first posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Stroke
Keywords: physical therapy; postural control; supra-postural task; stroke; motor control; contextual factors; variability
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Participants will receive physical therapist support to reduce postural sway while completing a precision aiming task in virtual reality, whether or not they require the support.
  Interventions: Behavioral: Physical therapist support
- Control Group (No Intervention): Participants will receive no physical therapist support while completing the task.

INTERVENTIONS:
Behavioral: Physical therapist support — Participants will receive physical therapist support to reduce postural sway variability while completing an upper limb precision aiming task in virtual reality.
  Arms: Experimental Group

SUMMARY:
The purpose of this study is to systematically determine the effect of unnecessary physical therapist assistance in individuals after stroke during the practice of an upper limb task on an individual's task performance and their underlying motor control patterns when learning (or re-learning) motor skills.

DETAILED DESCRIPTION:
Independent motor task performance is the most highly prioritized outcome of physical therapy for individuals with motor disability. Accordingly, a key priority for physical therapists in multiple practice settings is the advancement of functional motor independence. Therapists must determine when a patient requires assistance (e.g., verbal cues, physical support) to complete a motor task and when a patient is able to execute a motor skill with less assistance. If a therapist does not provide enough support, the patient is at risk for unsuccessful task performance. As such, therapists often default to providing a higher level of assistance.

An individual following stroke, for instance, may demonstrate an increased magnitude of postural sway while completing self-care activities at the sink. A therapist may decide to provide physical support for the patient to decrease sway variability, whether or not the patient requires this support to maintain performance. The motor control consequences of providing this assistance (thus constraining movement variability and providing fewer options for adapting movement) when assistance is actually not needed is unknown. The purpose of this study is to systematically determine the effect of unnecessary assistance during the practice of an upper limb task on functional performance and underlying motor control patterns when learning (or re-learning) motor skills in individuals with stroke. The insights gained from the current project will have the potential to improve the currently available physical therapy interventions for individuals with stroke.

The effects of unnecessary physical therapist support will be examined in terms of upper limb task performance, retention, and transfer, and in terms of the postural control supporting task performance. The study is currently planned for individuals with stroke. Participants will be required to maintain the position of a virtual laser within a target while standing. An experimental group will receive postural support (physical assistance to maintain upright posture) during a practice period in order to specifically determine the effect of postural support on upper limb task performance and postural sway patterns. Participants will also engage in a light finger force production transfer task to ascertain the influence of postural support on a different supra-postural task.

It is hypothesized that providing unnecessary assistance (and thus limiting independence) during practice of a novel motor task will result in (a) faster improvements in task performance but reduced retention and more limited transfer to another, similar task; and (b) reduced task- sensitive postural sway adjustments (measured in terms of both the quantity and temporal structure) during practice, at transfer, and at retention, reflecting reduced adaptability of postural patterns to task demands.

ELIGIBILITY:
Inclusion Criteria:

1. Between 45 and 80 years at time of consenting
2. Previous diagnosis of stroke for which they sought treatment (> 1 month prior to enrollment)
3. Able to communicate with investigators, follow a 2-step command and correctly answer consent comprehension questions
4. Independence or modified independence during ambulation (defined as the ability to ambulate with no physical assist and walk with an assistive device as needed) for at least 30 ft.
5. Score 0-3 on the Modified Rankin Scale, which indicates complete independence to moderate disability but able to walk without assistance.
6. Maintain standing balance for > 2 minutes with no physical support.
7. Maintain grasp of a handheld object with at least one hand.

Exclusion Criteria:

1. Limited language abilities, deafness, blindness, or serious motor impairment that outright prevents performance of the experimental tasks (e.g., severe lower extremity spasticity)
2. Pregnancy.
3. Pain with weightbearing > 4/10.
4. Inability to answer consent questions and follow simple 1-step commands.
5. Any other medical condition that would preclude the valid administration of the study measures, specifically seizure disorders or additional neurologic conditions beyond stroke.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2021-10-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cincinnati Center for Cognition, Action, and Perception, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Analytic code and other study materials may be shared on PI's Open Science Framework (OSF) page.
Supporting Information: Analytic Code
Time Frame: Within 6 months of study completion or after the primary manuscript from this study is accepted for publication and will likely remain available indefinitely
URL: https://osf.io/wq2rf/

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Limbs (Paretic/Non-Paretic)
Period: Overall Study
Arm/Group | Experimental Group | Control Group
Started | 13; 26 Limbs (Paretic/Non-Paretic) | 12; 24 Limbs (Paretic/Non-Paretic)
Completed | 11; 22 Limbs (Paretic/Non-Paretic) | 12; 24 Limbs (Paretic/Non-Paretic)
Not Completed | 2; 4 Limbs (Paretic/Non-Paretic) | 0; 0 Limbs (Paretic/Non-Paretic)
Not completed — Unable to complete experimental task | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Group | Control Group | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (4.3) | 50.8 (8.4) | 53.7 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 12 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 7 | 11
  White | 7 | 5 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Center of Pressure Path Length
Description: The amount of displacement of the location of the (resultant) vertical ground reaction force vector.
  Results only presented as the mean difference between groups, as only the paretic limb was used for this portion of the study. There are no results to report for the non-paretic limb.
Time Frame: 10 minutes of practice
Population: Difference between path length during practice.
Measure: Mean (Standard Error); unit: cm^2
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 11 | 12
cm^2 | 98.5 (17.5) | 156.1 (16.8)

2. Primary Outcome: Standard Deviation of Center of Pressure
Description: Variability of center of pressure trajectory.
Time Frame: After 10 minutes of practice
Population: Post-test results from when participants were aiming with each upper limb.
Measure: Mean (Standard Error); unit: cm
Groups:
- Experimental Group: Paretic Limb; Experimental Group: Non-Paretic Limb: Participants will receive physical therapist support to reduce postural sway while completing a precision aiming task in virtual reality, whether or not they require the support.
  Physical therapist support: Participants will receive physical therapist support to reduce postural sway variability while completing an upper limb precision aiming task in virtual reality.
- Control Group: Paretic Limb; Control Group Non-Paretic Limb: Participants will receive no physical therapist support while completing the task.
Arm/Group | Experimental Group: Paretic Limb | Control Group: Paretic Limb | Experimental Group: Non-Paretic Limb | Control Group Non-Paretic Limb
Number analyzed (Participants) | 11 | 12 | 11 | 12
cm | .70 (.06) | .53 (.05) | .69 (.04) | .53 (.04)

3. Primary Outcome: Percent Determinism of Postural Sway
Description: Quantifies the patterning, non-stationarity, and complexity of biological time series through the analysis of local recurrences in a reconstructed phase space. Highter values of percent determinism indicate more regularity in postural sway.
Time Frame: After 10 minutes of practice
Population: Post-test results
Measure: Mean (Standard Error); unit: percent determinism
Groups:
- Control Group: Non-Paretic Limb: Participants will receive no physical therapist support while completing the task.
Arm/Group | Experimental Group: Paretic Limb | Control Group: Paretic Limb | Experimental Group: Non-Paretic Limb | Control Group: Non-Paretic Limb
Number analyzed (Participants) | 11 | 12 | 11 | 12
percent determinism | .99 (.001) | .99 (.001) | .99 (.001) | .99 (.001)

4. Primary Outcome: Entropy (Sample Entropy)
Description: Evaluates the predictability of the next state of a system, given what is known about the current state of a system. Higher values of SampEn indicate less regularity; lower values indicate more regularity. Outcome measure reported as a ratio of anterior-posterior to medial-lateral SampEn values.
Time Frame: After 10 minutes of practice
Population: Post-test results
Measure: Mean (Standard Error); unit: ratio of AP:ML
Arm/Group | Experimental Group: Non-Paretic Limb | Control Group: Non-Paretic Limb | Experimental Group: Paretic Limb | Control Group: Paretic Limb
Number analyzed (Participants) | 11 | 12 | 11 | 12
ratio of AP:ML | 1.2 (.19) | 1.54 (.18) | 1.4 (.18) | 1.1 (.19)

5. Primary Outcome: Percent Correct
Description: Percent time on target.
Time Frame: After 10 minutes of practice
Population: Post-test results
Measure: Mean (Standard Error); unit: percentage of time on target
Arm/Group | Experimental Group: Paretic Limb | Control Group: Paretic Limb | Experimental Group: Non-Paretic Limb | Control Group: Non-Paretic Limb
Number analyzed (Participants) | 11 | 12 | 11 | 12
percentage of time on target | .66 (.08) | .74 (.06) | .95 (.01) | .91 (.01)

ADVERSE EVENTS:
Time Frame: No adverse events occurred during the study (1 hour, single session). Participants were only assessed for adverse events during the 1-hour single session
Description: There was no risk of death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal functions, or a congenital anomaly/birth defect by participating in this study.
Arm/Group | Experimental Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 0/11 | 0/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Group (N=11) | Control Group (N=12)
Fall (Musculoskeletal and connective tissue disorders) | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-07): https://cdn.clinicaltrials.gov/large-docs/27/NCT04856527/Prot_SAP_000.pdf